CLINICAL TRIAL: NCT01296178
Title: PROTOCOL FOR First Line TREATMENT ADAPTED TO RISK of Acute Myeloblastic Leukemia in Patients LESS THAN OR EQUAL TO 65 YEARS
Brief Title: PETHEMA-LMA10: Treatment of Acute Myeloblastic Leukemia (AML) in Patients Less Than or Equal to 65 Years
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PETHEMA-LMA10
Record Dates: First submitted 2011-02-09; First posted 2011-02-15 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Acute Myeloblastic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Idarubicin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: IDARUBICINE — Administration of chemotherapy induction
  Idarubicin IV Dose of 12 mg/m2/day days 1 to 3
Drug: ARA-C — ARA-C 200 mg/m2/day dose continuous infusion of IV days 1 to 7

SUMMARY:
Advances in the biological characterization of AML can now make a proper estimate of the risk of recurrence and likelihood of survival of different groups of patients according to the expression of different disease parameters. Karyotype, the molecular alterations affecting genes FLT3, NPM1 and CEBPA, minimal residual disease by flow cytometry and response to first induction cycle are variables that must be taken into consideration when planning the treatment of first line from a patient with AML.

This breakthrough in the field of biology has not resulted yet in the development of new drugs really effective in the treatment of AML. Therefore, the core of the treatment continue to rely on the use of traditional chemotherapy combined or not with allogeneic hematopoietic stem cell. Both treatments differ in their antileukemic efficacy, higher in aloTPH, as well as their toxicity and procedure-related mortality, increased also in the aloTPH. These aspects should be added that most candidates aloTPH patients lack an HLA identical sibling donor forcing the search for alternative sources and hematopoietic stem cell donors. These transplants alternative, but are not committed to their antileukemic efficacy, it does have implied a greater toxicity. Therefore, the ultimate effectiveness of these procedures depends largely on the proper selection of candidates for the same.

While there is broad agreement in terms of induction chemotherapy using a combination of cytarabine with anthracycline, the choice of chemotherapy regimen is controversial postremisión today. In the poor prognosis of itself involve the LMA, patients classified as "favorable group" are acceptable disease-free survival with consolidation schemes involving high-dose cytarabine. For other patients appear to be inappropriate to combine cytarabine with an anthracycline, at least one cycle of consolidation, and raise the option of allogeneic different depending on prognostic markers

DETAILED DESCRIPTION:
Primary objectives

1. Optimizing current treatment of AML based on the classification of patients into different risk groups according to parameters cytogenetic and molecular response to treatment and to analyze its effectiveness in terms of survival.
2. Apply a uniform treatment to individual patients according to previously defined prognostic groups.

Secondary Objectives

1. Correlate the different clinical and biological characteristics with response rates and patient outcomes.
2. Studying the role of minimal residual disease by molecular techniques in anticipation of relapse of AML

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML according to WHO criteria
* Previously untreated AML, including AML de novo,AML secondary to MDS or previous chemotherapy or radiotherapy
* No promyelocytic leukemia (no t (15, 17) or PML-RARa rearrangement and its variants)
* Age ≤ 65 years
* ECOG performance status 0-2
* Provide written informed consent
* Being able to comply with protocol procedures
* Not to be fertile or willing to use a method of birth control during treatment and until the end of it
* Adequate renal and hepatic function as follows, provided the changes, which would be not due to the disease: Total bilirubin < 1.5 x upper limit of normal (ULN) institutional and AST and ALT < 2.5 x ULN, and Serum creatinine < 2.5 mg / dL.
* Adequate cardiac function determined by at least 1 of the following:

Left ventricular ejection fraction (LVEF) > 40% measured by echocardiography in multiport scanner acquisition (MUGA) or isotope angiography, or Left ventricular fractional shortening > 22% measured in echocardiography

Exclusion Criteria:

* LPA diagnosis according to WHO criteria
* Previously untreated AML, except for the administration of hydroxyurea as a cytoreductive agent which itself is permitted
* AML secondary to chronic myeloproliferative syndrome
* Age> 65 years
* ECOG performance status> 2
* Absence of written informed consent
* Being unable to comply with protocol procedures
* Be fertile and not willing to use a method of birth control during treatment and until the end of it
* Hypersensitivity to any drug protocol
* Positive for HIV
* Abnormal liver and renal functions as indicated below, provided the changes, which would be not due to the disease: Total bilirubin> 1.5 x upper limit of normal (ULN) institutional and AST and ALT> 2.5 x ULN, and serum creatinine> 2.5 mg / dL
* Altered cardiac function determined by at least 1 of the following:

Left ventricular ejection fraction (LVEF) <40% measured by echocardiography in multiport scanner acquisition (MUGA) or isotope angiography, or Left ventricular fractional shortening <22% measured by echocardiography

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-12 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of survival months in treated AML patients less or equal to 65 years as a measure of survival time | 2 years
  Optimizing current treatment of AML based on the classification of patients into different risk groups according to parameters cytogenetic and molecular response to treatment and to analyze its effectiveness in terms of survival
Patients classification in prognostic groups | 2 years
  Patients classification in prognostic groups and aplication of individual treatments.

SECONDARY OUTCOMES:
Response rates | 2 years
  Correlate the different clinical and biological characteristics with response rates and patient outcomes
Determinate the minimal residual disease | 2 years
  Studying the role of minimal residual disease by molecular techniques in anticipation of relapse of AML

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital La Fe, Valencia, Spain